CLINICAL TRIAL: NCT01257464
Title: The Effects of the DPPIV Inhibitor Sitagliptin in Cystic Fibrosis-related Diabetes
Brief Title: Sitagliptin in Cystic Fibrosis-Related Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H08-02131
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
Keywords: CFRD; sitagliptin; cystic fibrosis-related diabetes; incretins; hyperglycemia; GIP; GLP-1
MeSH Terms: conditions — Cystic Fibrosis; Hyperglycemia | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100mg po one dose
  Other Names: Januvia, MK-0431, Dipeptidyl peptidase IV inhibitor (DPP-4 inhibitor)
  Arms: Sitagliptin
Drug: Placebo — Sugar pill po one dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the dipeptidyl peptidase IV (DPPIV) inhibitor sitagliptin is effective in the treatment of cystic fibrosis-related diabetes (CFRD). We hypothesize that sitagliptin will improve meal-stimulated insulin secretion.

DETAILED DESCRIPTION:
To date, no clinical trials have been conducted using the DPPIV inhibitor sitagliptin in cystic fibrosis-related diabetes. Cystic fibrosis-related diabetes is characterized initially by post-prandial hyperglycemia, with normal fasting sugars. As the disease progresses, fasting hyperglycemia develops. As sitagliptin augments post-prandial insulin release, while avoiding fasting hypoglycemia, it may be an alternative therapy for cystic fibrosis-related diabetes in individuals who do not yet require basal insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Cystic fibrosis-related diabetes with or without fasting hyperglycemia either untreated or using only pre-prandial repaglinide or pre-prandial bolus insulin therapy

Exclusion Criteria:

* Age under 19 years
* Use of basal insulin therapy
* Creatinine Clearance < 50 mL/min
* Active cystic fibrosis exacerbation
* Pregnancy
* Women of child-bearing age not using effective contraception
* Current or prior use of DPPIV inhibitor

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Insulin release | 180 minutes (during clamp)
  The study protocol is a iv-oral hyperglycemic glucose clamp. We will assess insulin release during the clamp, comparing placebo to sitagliptin.

SECONDARY OUTCOMES:
Incretin Response | 180 minutes (during clamp)
  We will assess incretin release [glucoagon-like peptide-1 (GLP-1), gastric inhibitory polypeptide(GIP)] during the glucose clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Gerontology & Diabetes Reserach Centre (ViTALITY), Vancouver, British Columbia, Canada